CLINICAL TRIAL: NCT00274261
Title: A Phase II/III Multicenter, Randomized, Double-masked, Study of the Safety and Contraceptive Efficacy of C31G Compared to Conceptrol®
Brief Title: Study of the Safety and Contraceptive Efficacy of C31G Compared to Conceptrol®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCN004; HHSN2752004033661
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy
Keywords: contraception
MeSH Terms: interventions — C 31G; Nonoxynol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): C31G vaginal gel contains 35mg (1% concentration) of C31G in 3.5 mL volume of gel
  Interventions: Drug: C31G
- B (Active Comparator): Conceptrol® Vaginal gel contains 100mg (4% concentration) of nonoxynol-9 (N-9) in 2.5 mL volume of gel.
  Interventions: Drug: nonoxynol-9 (N-9)

INTERVENTIONS:
Drug: C31G — The subject will insert one applicator of C31G prior to each episode of vaginal intercourse during her participation in the study.
  Arms: A
Drug: nonoxynol-9 (N-9) — The subject will insert one applicator of Conceptrol® vaginal gel (nonoxynol-9) prior to each episode of vaginal intercourse during her participation in the study.
  Arms: B

SUMMARY:
This is a multicenter, randomized, double-masked, controlled, phase III study of repeated use of C31G vaginal gel compared to Conceptrol® Vaginal Gel as the primary method of contraception over six months (183 days) and at least six cycles of use. In addition, there is an opportunity for subjects to continue with study treatment for up to twelve months (365 days) and twelve cycles of treatment upon completion of the first six months of treatment.

DETAILED DESCRIPTION:
Approximately 85% of American women (52 million) between the ages of 15 and 44 are sexually active . Approximately two-thirds or 38 million women use some form of birth control and/or STD prevention. With growing awareness of the risk of STDs, increasing numbers of women will require contraceptive methods that provide protection against STDs in addition to providing the basic contraceptive function. Currently there is no single, reasonably effective method to achieve both ends. Condoms, both male and female, present problems of acceptability for the partners of many at-risk women and, thus, cannot be considered an effective contraceptive and STD preventive for many people. A spermicide that also has the ability to prevent transmission of STDs would be a major advance, and of tremendous value to women worldwide.

C31G is an effective spermicide with in vitro activity equal to that of N-9 . C31G has been found to be a broad-spectrum antibacterial agent in vitro or in animals, active against both gram-positive and gram-negative organisms, including chlamydia, and a range of antibiotic resistant strains. It is also active against enveloped viruses including HIV and HSV. Thus, the primary objective of the study is to determine the contraceptive efficacy of C31G vaginal gel compared to Conceptrol® Vaginal Gel. The secondary objectives are to determine the safety and acceptability of the compounds with use over a period of six months or twelve months. Additional evaluations include the incidence of urinary tract infections (UTI), bacterial vaginosis (BV) and yeast vaginitis following the use of C31G vaginal gel compared to Conceptrol® Vaginal Gel.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must:

* Be healthy women, who are sexually active, at risk for pregnancy and desiring contraception.
* Be within the age range of 18 through 40 years inclusive.
* Be at low-risk for human immunodeficiency virus (HIV) or sexually transmitted disease (STD) infection and currently have a single sex partner (minimum 4 months) who is also at low-risk for HIV or STD.
* Have a negative urine pregnancy test prior to enrollment.
* Have normal cyclic menses with a usual length of 24 to 35 days over the last 2 cycles or at least one spontaneous, normal menstrual cycle (2 menses) since delivery, abortion, or after discontinuing hormonal contraception/hormonal therapy.
* Be willing to accept a risk of pregnancy.
* Be willing to engage in at least 4 acts of heterosexual vaginal intercourse per month for a period of 6 months.
* Be willing to be randomized to either study treatment.
* Be willing to only use the study product as the primary method of contraception over the course of the study with the exception of emergency contraception (EC), when indicated.
* Be capable of using the study product properly and agree to observe all study directions and requirements.
* Be willing to keep a diary to record coital information, product use information, information about the use of other vaginal products, and sign and symptom data of subject and partner.
* Agree not to participate in any other clinical trials during the course of the study.
* Be willing to give written informed consent to participate in the trial.

Exclusion Criteria:

Potential subjects must not:

* Have a history of allergy or sensitivity to spermicides or products containing N-9.
* Have had 3 or more urinary tract infections (UTI) in the past year.
* Have UTI by urine culture or symptomatic yeast vaginitis or symptomatic bacterial vaginosis diagnosed by wet mount unless treated and proof of cure is documented.
* Be pregnant, have a suspected pregnancy or desire to become pregnant during the course of the study.
* Have a history of infertility or of conditions that may lead to infertility, without subsequent intrauterine pregnancy.
* Have any contraindications to pregnancy (medical condition) or chronic use of category D or X medications.
* Have had more than one sexual partner in the last 4 months.
* Have shared injection drug needles within the past 12 months.
* Have or have been suspected to have HIV infection.
* Have been diagnosed with genital herpes simplex virus (HSV), with the first occurrence (initial episode) within three months prior to screening.
* Have 3 or more outbreaks of HSV within the last year.
* Have been diagnosed with any other STDs (including trichomonas) in the 6 months prior to the screening visit (with the exception of Human Papilloma Virus [HPV]).
* Be lactating or breastfeeding.
* Have any clinically significant abnormal vaginal bleeding or spotting within the month prior to screening.
* Have any clinically significant abnormal finding on pelvic examination or baseline labs, which in the view of the investigator, precludes her from participating in the trial.
* Have clinically significant signs of vaginal or cervical irritation on pelvic examination.
* Have had vaginal or cervical biopsy or vaginal surgery within 3 months prior to screening.
* Have used vaginal or systemic antibiotics or antifungals within 14 days prior to screening or randomization.
* Have had a Depo-Provera® injection in the 10 months prior to enrollment.
* Have an abnormal Pap smear with high grade squamous intraepithelial lesion (HSIL), atypical glandular cells (AGC) or ASC-H (atypical squamous cells, cannot exclude HSIL) within the last 12 months.
* Have an abnormal Pap smear with low-grade squamous intraepithelial lesion (LSIL) or ASCUS-HPV HR positive unless resolved by colposcopy.
* Have a Cervical Intraepithelial Neoplasia (CIN) diagnosis by biopsy within the last 12 months.
* Have a history or a current diagnosis of cervical cancer.
* Consume (on average) greater than three drinks of an alcoholic beverage per day.
* Have a past history (within twelve months) or current history of drug abuse [recreational, prescription or over-the-counter (OTC)].
* Have taken an investigational drug or used an investigational device within the past 30 days.
* Have previously participated in or completed this study or any other phase III study of C31G.
* Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1565 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Blithe, Ph.D., Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (15):
- United States (15):
  - California Family Health Council, Berkeley, California
  - California Family Health Council, Los Angeles, California
  - University of Colorado - Advanced reproductive Medicine, Aurora, Colorado
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Bay State Medical Center, Springfield, Massachusetts
  - New York University, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland MacDonald Women's Hospital, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - U.T. Southwestern Medical Center, Dallas, Texas
  - Jones Institute of Reproductive Medicine, EVMS, Norfolk, Virginia

REFERENCES:
- [Derived] Burke AE, Barnhart K, Jensen JT, Creinin MD, Walsh TL, Wan LS, Westhoff C, Thomas M, Archer D, Wu H, Liu J, Schlaff W, Carr BR, Blithe D. Contraceptive efficacy, acceptability, and safety of C31G and nonoxynol-9 spermicidal gels: a randomized controlled trial. Obstet Gynecol. 2010 Dec;116(6):1265-1273. doi: 10.1097/AOG.0b013e3181fc3b1a. PMID 21099590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female subjects were screened and enrolled at 15 sites in the US.
Groups:
- C31G: C31G vaginal gel contains 35mg (1% concentration) of C31G in 3.5 mL volume of gel
- Conceptrol: Conceptrol® Vaginal gel contains 100mg (4% concentration) of nonoxynol-9 (N-9) in 2.5mL volume of gel.
Period: Overall Study
Arm/Group | C31G | Conceptrol
Started | 932 | 633
Completed | 443 | 296
Not Completed | 489 | 337
Not completed — Adverse Event | 19 | 11
Not completed — Pregnancy | 114 | 83
Not completed — Withdrawal by Subject | 179 | 126
Not completed — Protocol Violation | 71 | 42
Not completed — Lost to Follow-up | 106 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C31G | Conceptrol | Total
Number analyzed (Participants) | 932 | 633 | 1565
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 932 | 633 | 1565
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.58) | 28.3 (5.90) | 28.2 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 932 | 633 | 1565
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 932 | 633 | 1565

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Probability of Typical-use 6 Month (183 Days) Pregnancy.
Description: Number of pregnancies in women using C31G gel for 6 months (183 days) compared to women using Conceptrol gel for the same time frame.
Time Frame: 6 months
Population: Modified Intent-To-Treat (MITT): ITT subjects whose diaries indicated they had at least one episode of coitus while using the assigned study product (also referred as "Typical-Use") and for whom there is at least one report of pregnancy status.
Measure: Number (95% Confidence Interval); unit: 6 month probability of pregnancy
Arm/Group | C31G | Conceptrol
Number analyzed (Participants) | 827 | 555
6 month probability of pregnancy | 0.12 [0.093 to 0.147] | 0.12 [0.087 to 0.153]

2. Secondary Outcome: Incidence of Adverse Events.
Description: Evaluated by comparing the incidence of Adverse Events (AEs) among subjects using their assigned treatment for at least one day.
Time Frame: duration of the study - through 6 month or 12 months of use
Measure: Count of Participants; unit: Participants
Groups:
- C31G Vaginal Gel: C31G vaginal gel contains 35mg (1% concentration) of C31G in 3.5 mL volume of gel
  C31G: The subject will insert one applicator of C31G prior to each episode of vaginal intercourse during her participation in the study.
- Conceptrol® Vaginal Gel: Conceptrol® Vaginal gel contains 100mg (4% concentration) of nonoxynol-9 (N-9) in 2.5 mL volume of gel.
  nonoxynol-9 (N-9): The subject will insert one applicator of Conceptrol® vaginal gel (nonoxynol-9) prior to each episode of vaginal intercourse during her participation in the study.
Arm/Group | C31G Vaginal Gel | Conceptrol® Vaginal Gel
Number analyzed (Participants) | 932 | 633
Participants | 617 | 434

ADVERSE EVENTS:
Description: The overall safety population includes only subjects that actually used the product at least once totalling 1396.
Arm/Group | C31G | Conceptrol
Serious Adverse Events (participants affected / at risk) | 10/836 | 12/560
Other Adverse Events (participants affected / at risk) | 617/836 | 434/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C31G (N=836) | Conceptrol (N=560)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis escherichia coli (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermoid Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Cyst Ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningitis viral (Nervous system disorders) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Kidney Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C31G (N=836) | Conceptrol (N=560)
Nasopharygitis (Infections and infestations) | 130 | 92
Vaginitis bacterial (Infections and infestations) | 100 | 73
Vaginal mycosis (Infections and infestations) | 87 | 70
Headache (Nervous system disorders) | 79 | 63
Urinary tract infection (Infections and infestations) | 79 | 59
Metrorrhagia (Reproductive system and breast disorders) | 69 | 55
Menstrual cycle prolonged (Reproductive system and breast disorders) | 57 | 41
Menstruation irregular (Reproductive system and breast disorders) | 56 | 41
Influenza (Infections and infestations) | 57 | 35
Dysmenorrhoea (Reproductive system and breast disorders) | 49 | 37
Genital pruritus female (Reproductive system and breast disorders) | 30 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 25
Oligomenorrhoea (Reproductive system and breast disorders) | 38 | 19
Smear cervix abnormal (Investigations) | 32 | 24
Pharyngolaryngeal pain (Gastrointestinal disorders) | 32 | 20
Toothache (Gastrointestinal disorders) | 30 | 12
Abdominal pain upper (Gastrointestinal disorders) | 21 | 16
Upper respiratory tract infection (Infections and infestations) | 18 | 15
Nausea (Gastrointestinal disorders) | 18 | 12
Vaginal burning sensation (Reproductive system and breast disorders) | 16 | 13
Sinusitis (Infections and infestations) | 14 | 14
Vulvovaginal discomfort (Reproductive system and breast disorders) | 12 | 16
Vaginal odor (Reproductive system and breast disorders) | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other